CLINICAL TRIAL: NCT04256057
Title: Effect of Intraoperative Magnesium Infusion on Postoperative Pain and Cognitive Function After Pelvi-abdominal Surgeries :an Observational Study
Brief Title: Effect of Intraoperative Magnesium Infusion on Postoperative Pain and Cognitive Function
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Samaa Rashwan, Samaa Abou Alkassem Rashwan, Beni-Suef University
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: faculty of medicine Beni-Suef
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: the Effect of Intraoperative Magnesium Infusion on Postoperative Cognitive Functions in Adult Patients After Elective Pelvi-abdominal Surgeries
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- magnesium sulphate (Other): After the induction of anesthesia, a loading dose of magnesium sulfate 50mg/kg in 100mL of isotonic saline as within 5 to 10 minutes followed by a maintenance dose of 10 mg/kg/hr up to the end of surgery
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — After the induction of anesthesia, a loading dose of magnesium sulfate 50mg/kg in 100mL of isotonic saline as within 5 to 10 minutes(23) followed by a maintenance dose of 10 mg/kg/hr up to the end of surgery

SUMMARY:
The aimof this study is to observe the effect of intraoperative magnesium infusion on peri-operative pain and postoperative cognitive functions in adult patients after elective pelvi-abdominal surgeries.

DETAILED DESCRIPTION:
This study will be conducted at Beni-Suef University Hospital after approval of the anesthesiology, surgical ICU and pain management department, and the local ethics and research committee, and obtaining written informed consents from the patients .

The inclusion criteria:

1. Male and female patients (age 20-60 years)
2. American Society of Anesthesiology(ASA) physical status I-II
3. Patients scheduled for elective pelvi-abdominal surgeries

The Exclusion criteria

1. Patients having significant cardiovascular (cardiomyopathy or moderate to severe valvular heart lesion) , significant hepatic disease (Child-Pugh score B or C ), renal or CNS disease
2. Patients with uncontrolled hypertension or diabetes
3. History of hypersensitivity to the drugs to be used
4. Control MMSE score ≤23
5. Women who are pregnant or breastfeeding
6. Patients taking Ca2+ channel blockers, opioids, antidepressants, or antipsychotics or alcohol
7. Patients having difficulty understanding , vision or hearing problems or CNS disorder as parkinson's disease .
8. Morbidly obese patients with a body mass index of >40
9. Patients who refused to be involved within the scope of the research. Management of the patients in the operation room All patients will be informed about the tests and written informed consent will be obtained from each of them. The MMSE will be applied. After arrival to the operation theater the monitors will be applied including will be applied including 5 leads ECG, non invasive arterial blood pressure and pulse oximetry. Urinary catheter will be inserted for urine output monitoring. Train of four (TOF) monitoring and Bispectral index (BIS) monitoring will be done in order to evaluate the depth of hypnosis (A-2000 Bispectral Index, Aspect Medical Systems, the Netherlands).

Following 100% oxygen of 5 L/min for 3 min, 1% lidocaine at 0.5 mg/kg will be given intravenously in order to prevent potential injection pain due to propofol and to suppress hemodynamic response to endotracheal intubation. Propofol 2 mg/kg, midazolam 0.03 mg/kg, fentanyl 3μg/kg and 0.6 mg /kg atracurium will be given followed by intubation and Mechanical ventilation with 6 mL/kg tidal volume and a frequency of 8-12/min with total of 4 L/min in 40% O2 air mixture to keep EtCO2 between 36 and 40 mmHg. Anesthesia will be maintained using oxygen and 1-1.5 minimum alveolar concentration (MAC) of isoflurane.

After the induction of anesthesia, a loading dose of magnesium sulfate 50mg/kg in 100mL of isotonic saline as within 5 to 10 minutes followed by a maintenance dose of 10 mg/kg/hr up to the end of surgery .24 In case of a patient with hypotension (mean arterial pressure ˂55 mmHg), 5 mg ephedrine will be injected so that the mean arterial pressure could reach higher than 55 mm Hg. If arrhythmia occured in any of the patients during operation, proper treatment will be be performed and the patient will be excluded from the study. The magnesium sulphate and anaesthetic agent infusions will be discontinued at skin closure. The relaxant effect of magnesium sulfate will be considered so train of four (TOF) monitoring will be used to monitor the muscle relaxation during the surgery and patients will be extubated at the end of the operation based on the TOF > 0.9 to ensure the complete reversal of relaxants by neostigmin.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients (age 20-60 years)
2. American Society of Anesthesiology(ASA) physical status I-II
3. Patients scheduled for elective pelvi-abdominal surgeries

Exclusion Criteria:

1. Patients having significant cardiovascular (cardiomyopathy or moderate to severe valvular heart lesion) , significant hepatic disease (Child-Pugh score B or C ), renal or CNS disease
2. Patients with uncontrolled hypertension or diabetes
3. History of hypersensitivity to the drugs to be used
4. Control MMSE score ≤23
5. Women who are pregnant or breastfeeding
6. Patients taking Ca2+ channel blockers, opioids, antidepressants, or antipsychotics or alcohol
7. Patients having difficulty understanding , vision or hearing problems or CNS disorder as parkinson's disease .
8. Morbidly obese patients with a body mass index of >40
9. Patients who refused to be involved within the scope of the research.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-04-15 (Estimated)

PRIMARY OUTCOMES:
magnesium infusion on postoperative cognitive functions in adult patients after elective pelvi-abdominal surgeries. | the observation will be for 24 hours
  After the induction of anesthesia, a loading dose of magnesium sulfate 50mg/kg in 100mL of isotonic saline as within 5 to 10 minutes(23) followed by a maintenance dose of 10 mg/kg/hr up to the end of surgery

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Beni-Suef University Hospital, Banī Suwayf
  - Faculty of Medicine, Beni-SuefUniversity, Giza
  - Faculty of Medicine,Beni-Suef University, Giza

IPD SHARING:
Plan to Share IPD: No